CLINICAL TRIAL: NCT01180140
Title: Use of Seamguard to Prevent Digestive Leak and Bleeding on Lineal Stapled Anastomoses: a Prospective Randomized Clinical Trial
Brief Title: Use of Seamguard to Prevent Leak and Bleeding in Gastrointestinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario de Canarias (Other)
Collaborators: Unidad mixta de Investigación HUC-ULL (Unknown); University of La Laguna (Other)
Responsible Party: Mª Cruz Correa Flores, HUC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Seamguard Study
Record Dates: First submitted 2010-07-18; First posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Leak on Lineal Stapled Anastomoses; Bleeding on Lineal Stapled Anastomoses
Keywords: Seamguard; staple-line reinforcement; leak; bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): without seamguard
- 2 (Experimental): with seamguard
  Interventions: Device: Seamguard

INTERVENTIONS:
Device: Seamguard — GORE SEAMGUARD® Bioabsorbable Staple Line Reinforcement is specifically engineered to reduce the incidence of perioperative leaks and bleeding in a variety of open and minimally invasive surgeries. Then, after six months, it is completely absorbed eliminating the risk of a prolonged inflammatory response.
  Arms: 2

SUMMARY:
The purpose of this study is to determinate the utility of staple-line reinforcement on lineal gastrointestinal anastomoses.

Hypothesis: Seamguard device will decrease the incidence of leak and bleeding in digestive lineal stapled anastomoses.

ELIGIBILITY:
Inclusion Criteria:

* All patients who will need a lineal stapled anastomoses (colon cancer in cecum, for example)

Exclusion Criteria:

* circular anastomoses
* bariatric surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2006-03; Primary Completion 2009-08 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz de Tenerife, Spain